CLINICAL TRIAL: NCT05980351
Title: Effect of Exercise Program on Quality of Life and Stress in Children Undergoing Hemodialysis
Brief Title: Exercise Program on Quality of Life and Stress in Children Undergoing Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Hassan Khalf allah, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Exercise on QOL and stress
Record Dates: First submitted 2023-07-29; First posted 2023-08-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Quality of Life
Keywords: Exercise; Quality of Life; Stress; Hemodialysis children
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): This group will receive exercise program
  Interventions: Other: exercise
- Control group (No Intervention): This group will receive routine hospital care

INTERVENTIONS:
Other: exercise — The children will receive exercise program(stretching exercise,range of motion exercise and isometric exercise)
  Arms: Study group

SUMMARY:
Despite the benefits of physical exercises among children with chronic illness, the children avoid to engage in different physical activities because their parent and the child also were faired to happen any complication to child. The lack of activity and sedentary life style among these children result in reduced quality of life in addition to behavioral and social problems and finally become independent in most of activities of daily living. Therefore, the primary aim of this study will to practice and teach the children exercise programs in order to improve the quality of life and reduce stress in children undergoing hemodialysis. Therefore aim of this study is to: Determine the effect of exercise program on quality of life and stress in children undergoing hemodialysis.

DETAILED DESCRIPTION:
* The researcher will go to hospital and will take all children that present in hemodialysis unit, then will make random assignment of children to study or control group .The control group will receive routine care while the study group will receive exercise program.
* The exercise program will conduct three days per week giving an interval of 24 hours between sessions. In the first hour the child not make any activity, then first 20 min from second hour of hemodialysis the child will receive stretching exercise, first 20 min from third hour the child will receive range of motion exercise finally first 20 min from forth hour the child will practice isometric exercise.
* This procedure will continue for 2 months and the end of time the research will make posttest for both groups. The intensity for resistance training will determined individually. Depending up on the child exercise tolerance, each set will performed 10 gradually increase to 15 repetitions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 6-18years with chronic renal failure.

  * All children are stable on dialysis for 2 months (Blood pressure under medical control and stable blood sugar).
  * All children are free from lower extremity graft and any lower limb pathology.
  * Children do not take exercise in 6 months before treatment.
  * Willing to participate in the study and attend the exercise schedule.
  * Children able to follow verbal commands.

Exclusion Criteria:

* Children with physical disabilities.
* Children on tranquilizers or sedative medications.
* Children with a femoral dialysis catheter& internal jugular vein catheter

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Children Quality Of Life | After 2 months
  Health Related Quality Of Life (HRQOL): Will use to measure children quality of life which includes the four domains (physical, emotional, social and school performance), each domain consists of 5 questions. Each question will earn score from (0-4) according to their answer as the following:
  4 means= never have a problem 3 means= almost never a problem 2 means= sometimes a problem
  1 means= it is often a problem 0 means = almost always a problem
Stress | After 2 months
  Tool (3): Perceived Stress Scale The Perceived Stress Scale (PSS) is a classic stress assessment instrument. This tool, helping the investigators to understands how different situations affect participants feelings and perceived stress. The questions in this scale ask about participants feelings and thoughts. In each case, the child will be asked to indicate how often felt or thought a certain way.
  This scale consisted of 10 questions; each question will earn score from (0-4) according to their answer as the following:
  4 means= very often 3 means= fairly often 2 means= sometimes
  1 means= almost never 0 means = never Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.

IPD SHARING:
Plan to Share IPD: No